CLINICAL TRIAL: NCT05840406
Title: Effect of a Transversus Abdominis Plane Block on Operative Wound Healing, Stress, and Immune Response After a Cesarean Delivery
Brief Title: Effect of a Transversus Abdominis Plane Block on Wound Healing, Stress, and Immune Response After a Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Mirta Ciglar, MD, Principal Investigator, University Hospital Sestre Milosrdnice
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 003-06/22-03/007
Record Dates: First submitted 2023-04-14; First posted 2023-05-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain; Cesarean Section; Wound Heal
Keywords: Cesarean section; Wound healing; Nerve block; Cortisol; Immune response
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Levobupivacaine; Dexmedetomidine; Tramadol; Ketoprofen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Prospective single-blind randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomly allocated to either a group SA receiving the standard postoperative analgesia or groups receiving the TAP block with levobupivacaine (group L) or levobupivacaine with the addition of dexmedetomidine (group D). The allocation sequence will be generated by a random number table. After signing an informed consent, participants and an anesthesiologist performing the TAP block will be informed about patients' group allocation. An independent observer, who will not know which group the participant belongs to, will assess wound healing using the standardized REEDA scale 72 hours after the cesarean delivery. The same independent observer will assess every participant at 4, 8, 12, 18, 24, and 72 hours after surgery for pain by using the pain numerical rating scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group SA (Active Comparator): No TAP block applied.
  Interventions: Drug: Postoperative pain management with acetaminophen; Drug: Postoperative pain management with tramadol; Drug: Postoperative pain management with ketoprofen; Drug: Postoperative pain management with ibuprofen
- Group L (Experimental): Ultrasound-guided bilateral TAP block (in-plane technique) will be performed in this group. Levobupivacaine 0.25 % 20 ml will be administered in the block on each side.
  Interventions: Drug: Postoperative pain management with acetaminophen; Procedure: Bilateral TAP Block with levobupivacaine; Drug: Postoperative pain management with tramadol; Drug: Postoperative pain management with ketoprofen; Drug: Postoperative pain management with ibuprofen
- Group D (Experimental): Ultrasound-guided bilateral TAP block (in-plane technique) will be performed in this group. Levobupivacaine 0.25 % 20 ml + dexmedetomidine 0,5 μg/kg will be administered in the block on each side.
  Interventions: Drug: Postoperative pain management with acetaminophen; Procedure: Bilateral TAP Block with levobupivacaine and dexmedetomidine; Drug: Postoperative pain management with tramadol; Drug: Postoperative pain management with ketoprofen; Drug: Postoperative pain management with ibuprofen

INTERVENTIONS:
Drug: Postoperative pain management with acetaminophen — During the 24 hours postoperatively, participants will receive 1 g acetaminophen intravenously (i.v.) three times a day. On the second and third postoperative days, participants will receive 1g acetaminophen per os three times a day.
Procedure: Bilateral TAP Block with levobupivacaine — Ultrasound-guided bilateral TAP block will be performed, and 20 ml of 0,25 % levobupivacaine will be administered to the participant on each side.
  Arms: Group L
Procedure: Bilateral TAP Block with levobupivacaine and dexmedetomidine — Ultrasound-guided bilateral TAP block will be performed, and 20 ml of 0,25 % levobupivacaine with the addition of 0,5 μg/kg dexmedetomidine will be administered to the participant on each side.
  Arms: Group D
Drug: Postoperative pain management with tramadol — During the 24 hours postoperatively, participants will receive 500 mg tramadol + 500 ml 0,9% NaCl i.v. continuously 30ml/h.
Drug: Postoperative pain management with ketoprofen — During the 24 hours postoperatively, participants will receive 100 mg ketoprofen + 100 ml of 0,9% NaCl i.v. twice a day. The first dose will be administered in the theatre at the end of the surgical procedure.
Drug: Postoperative pain management with ibuprofen — On the second and third postoperative days, participants will receive 600 mg ibuprofen per os three times a day.

SUMMARY:
The primary purpose of this study is to determine whether the addition of a TAP block to standard analgesia after the cesarean delivery will impact postoperative wound healing and attenuate postoperative stress and immune response.

Random allocation of participants in 3 groups: group SA (standard analgesia), group L (TAP block with levobupivacaine), and group D (TAP block with levobupivacaine + dexmedetomidine). All participants will undergo elective cesarean section through Pfannestiel incision under spinal anesthesia. They will receive standard postoperative pain management with acetaminophen, nonsteroidal anti-inflammatory drugs, and tramadol. Groups L and D will additionally receive bilateral ultrasound-guided TAP block with 20 ml 0,25% levobupivacaine or with 20 ml 0,25% levobupivacaine with the addition of 0,5 μg/kg dexmedetomidine. TAP block will be performed in the theatre immediately after the cesarean delivery.

Venous blood samples will be collected before the surgery and on the third postoperative day. Complete blood count and serum cortisol levels will be measured. REEDA scale will be used for assessing wound healing.

DETAILED DESCRIPTION:
Introduction. Cesarean section is one of the world's most frequently performed surgical procedures. It is often accompanied by severe postoperative pain that leads to a complex immune and stress response in the body. Neutrophil to lymphocyte ratio (NLR) and platelet to lymphocyte ratio (PLR) are reliable and readily available markers of immune response to various infectious and non-infectious stimuli. Elevated NLR and PLR values are predictive in the early detection of wound infection after cesarean section. Wound healing involves three stages: inflammation, proliferation, and remodeling. REEDA scale is a valid tool for assessing obstetric wound healing. Many factors can affect the wound-healing process. Consistent overlap between pain-related dysregulation of neuroendocrine and immune function and the aspects of the neuroendocrine and immune function shown to be critical in wound healing suggests that pain may play a role in delayed wound healing. Therefore, it is reasonable to assume that better postoperative analgesia could positively affect wound healing. According to previous research, the transversus abdominis plane (TAP) block significantly reduces pain and cortisol, epinephrine, and norepinephrine levels after cesarean section. The addition of dexmedetomidine to the local anesthetic in the TAP block has a more pronounced analgesic effect and prolongs the duration of analgesia. The investigators have found only one study that demonstrates that adding a TAP block to standard analgesia positively affects wound healing after cesarean delivery. In the literature search, investigators did not find any clinical study that has been carried out to see the influence of the addition of dexmedetomidine in TAP block on wound healing, stress response, and immune response after cesarean delivery.

We hypothesize that the use of bilateral transversus abdominis plane block after cesarean delivery will lead to lower values of the REEDA scale and attenuated stress and immune response of the patient compared to standard analgesia, where the addition of dexmedetomidine to levobupivacaine will have a more pronounced effect compared to TAP block with levobupivacaine.

Patients and methods: This prospective, randomized study will be conducted in the Department of Anesthesiology, Intensive Care Medicine and Pain Management and the Department of Gynecology and Obstetrics in the Sestre Milosrdnice University Hospital Center. A total of 120 participants will be included in the study.

The group size was obtained by power analysis. For each variable, the sample size required for cross-comparisons of the arithmetic means of the three groups was calculated using a two-tailed t-test with the power of the test β = 85%, and the level of statistical significance for each test, α = 1.667%. Standard deviations and expected differences in the arithmetic means of the examined groups were taken from the published literature. (2:24-26). The largest estimated sample size for the investigated variables is 35 subjects per group.

After the written and signed approval of the patients, they will be randomly allocated to either a control group that receives the standard postoperative analgesia (group SA) or groups that further receive the TAP block with levobupivacaine (group L), with and without the addition of dexmedetomidine (group D). All the participants will undergo elective cesarean delivery under spinal anesthesia. The classic cesarean section technique described by Pfannenstiel and Kerr technique will be performed on all the participants. The spinal anesthesia will be performed with an atraumatic spinal needle by applying height- and weight-adjusted dose of hyperbaric bupivacaine and 25 μg fentanyl intrathecally. All the participants will receive standard postoperative analgesia according to the Acute Pain Service Sestre Milosrdnice University Hospital Center (acetaminophen, tramadol, and nonsteroidal anti-inflammatory drugs). Group L and group D will additionally receive a bilateral TAP block. 20 ml of 0,25 % levobupivacaine will be administered on each side to the participants in group L and 20 ml of 0,25 % levobupivacaine with the addition of 0,5 μg/kg dexmedetomidine will be administered on each side to the participants in group D. TAP block will be performed under sterile conditions. The high-frequency linear probe will be placed transversally in the medial axillary line, and the three layers of abdominal muscles will be visualized. A 22G echogenic needle for peripheral nerve blocks will be used to inject the mixed solution in the plane between the transversus abdominis and internal oblique muscles.

Venous blood samples will be collected the day before the surgery, at 7 a.m. on the day of surgery, and at 7 a.m. on the third postoperative day. Complete blood count and serum cortisol levels will be measured. An independent observer will assess wound healing using the standardized Redness, edema, ecchymosis, discharge, and approximation (REEDA) scale 72 hours after the cesarean delivery.

Statistical analysis: The collected data for each variable will be summarized and analyzed depending on the normality of the distribution, which will be tested with the Shapiro-Wilk test. In the case of a normal distribution, the measured values will be summarized by the arithmetic mean and standard deviation. The effects of the treatment will be tested with a mixed model in which the measured value will be the dependent variable. In case of deviation from the normal distribution, the measured values will be summarized by the meridian and the first and third quartiles. Before the analysis with the mixed model they will be transformed by the inverse transformation of the ranks into the standard normal function. The calculated p-values will be considered statistically significant if they are less than 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for the elective cesarean section through Pfannenstiel incision under spinal anesthesia
* Age >18
* American Society of Anesthesiologists (ASA) physical status II
* Body mass index < 40 mg/kg²
* >35 gestational weeks

Exclusion Criteria:

* participant's refusal to participate in the study
* ASA physical status >II
* emergency cesarean section
* twin or triplets pregnancy
* history of allergy to the local anesthetic or any other drug used in this study (dexmedetomidine, acetaminophen, tramadol, nonsteroidal anti-inflammatory drugs)
* contraindications for spinal anesthesia or TAP block

Drop out from the study:

* the change in anesthetic technique from spinal to the general anesthesia
* the need for the blood transfusion
* acute mastitis, puerperal endometritis, and/or wound infection developed in the first 72 hours postoperatively
* failed TAP block

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Wound healing | 72 hours after the surgery
  Wound healing will be assessed 72 hours after cesarean delivery using a standardized REEDA scale. REEDA includes five factors associated with the healing of an incision: redness, edema, ecchymosis, discharge, and approximation of the two edges of the wound, each receiving a score between 0-3, with a higher score indicating a greater level of tissue trauma and less healed wound compared to lower scores.
Measure the stress response (serum cortisol) | up to 72 hours
  Venous blood samples will be collected at 7 a.m. on the day of surgery and at 7 a.m. on the 3rd postoperative day. Serum cortisol levels will be measured by using electrochemiluminescence immunoassay (ECLIA).
Measure immune response (neutrophil to lymphocyte ratio) | up to 72 hours
  The neutrophil to lymphocyte ratio will be calculated as a simple ratio between absolute neutrophil and lymphocyte counts measured in peripheral blood. Venous blood samples will be collected the day before the surgery at the admission and at 7 a.m. on the third postoperative day.
Measure immune response (platelet to lymphocyte ratio) | up to 72 hours
  The platelet to lymphocyte ratio will be calculated as a simple ratio between absolute platelet and lymphocyte counts measured in peripheral blood. Venous blood samples will be collected the day before the surgery at the admission and at 7 a.m. on the third postoperative day.

SECONDARY OUTCOMES:
Postoperative pain score | 4, 8, 12, 18, 24, and 72 hours after surgery
  A Numeric Rating Scale will measure pain at rest and on movement. The numeric Rating Scale will be from 0 to 10, where 0 is no pain, and 10 is the most severe pain. Pain will be assessed for each participant at 4, 8, 12, 18, 24, and 72 hours after surgery.
Quality of recovery | 24 hours after the surgery
  The quality of recovery will be measured by the Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool 24 hours after the surgery. ObsQoR-10© is a 10-item, participant-reported scoring tool that assesses postpartum recovery. It consists of 2 parts. In the first part, the subject self-evaluates the intensity of the four listed symptoms on a vertical visual-analog scale. The end points are marked with 0 - no symptoms and 10 - the worst possible intensity of symptoms. The second part consists of 6 questions assessing recovery in the last 24 hours, which the respondent also evaluates with a vertical visual-analog scale where the end points are marked with 0 - never and 10 - always. Possible scores range from 0 to 100, with a higher score indicating better postpartum recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Mirta Ciglar, MD, Principal Investigator — University Hospital Center Sestre Milosrdnice
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavand'homme P. Postoperative cesarean pain: real but is it preventable? Curr Opin Anaesthesiol. 2018 Jun;31(3):262-267. doi: 10.1097/ACO.0000000000000585. PMID 29521684
- [Background] Ernawati E, Amirah A, Sumartono C, Aditiawarman A. Comparison of Post-Caesarean Section Wound Healing Methods Based on Reeda Scale and Platelet Lymphocyte Ratio. Syst Rev Pharm. 2020;11(7):5. doi:10.31838/srp.2020.7.49
- [Background] Rotem R, Erenberg M, Rottenstreich M, Segal D, Yohay Z, Idan I, Yohay D, Weintraub AY. Early prediction of post cesarean section infection using simple hematological biomarkers: A case control study. Eur J Obstet Gynecol Reprod Biol. 2020 Feb;245:84-88. doi: 10.1016/j.ejogrb.2019.12.009. Epub 2019 Dec 23. PMID 31884150
- [Background] Hughes O, MacQuhae F, Rakosi A, Herskovitz I, Kirsner RS. Stress and wound healing. U: França K, Jafferany M, ur. Stress and skin disorders: Basic and clinical aspects. Cham: Springer; 2017. P. 185-207.
- [Background] Childs C, Sandy-Hodgetts K, Broad C, Cooper R, Manresa M, Verdu-Soriano J. Risk, Prevention and Management of Complications After Vaginal and Caesarean Section Birth. J Wound Care. 2020 Nov 1;29(Sup11a):S1-S48. doi: 10.12968/jowc.2020.29.Sup11a.S1. No abstract available. PMID 33170077
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Liu R, Qin H, Wang M, Li K, Zhao G. Transversus abdominis plane block with general anesthesia blunts the perioperative stress response in patients undergoing radical gastrectomy. BMC Anesthesiol. 2019 Nov 7;19(1):205. doi: 10.1186/s12871-019-0861-0. PMID 31699052
- [Background] Varshney A, Prabhu M, Periyadka B, Nanjundegowda DC, Rao A. Transversus abdominis plane (TAP) block with levobupivacaine versus levobupivacaine with dexmedetomidine for postoperative analgesia following cesarean delivery. J Anaesthesiol Clin Pharmacol. 2019 Apr-Jun;35(2):161-164. doi: 10.4103/joacp.JOACP_372_17. PMID 31303702
- [Background] Sun Q, Liu S, Wu H, Ma H, Liu W, Fang M, Liu K, Pan Z. Dexmedetomidine as an Adjuvant to Local Anesthetics in Transversus Abdominis Plane Block: A Systematic Review and Meta-analysis. Clin J Pain. 2019 Apr;35(4):375-384. doi: 10.1097/AJP.0000000000000671. PMID 30475260
- [Background] Surhonne N, Hebri C, Kannan S, Duggappa DR, Rs RR, Mapari CG. The effect of anesthetic techniques on neutrophil to lymphocyte ratio in patients undergoing infraumbilical surgeries. Korean J Anesthesiol. 2019 Oct;72(5):458-465. doi: 10.4097/kja.d.19.00022. Epub 2019 May 17. PMID 31096728
- [Background] Kiriakopoulos N, Grigoriadis S, Maziotis E, Philippou A, Rapani A, Giannelou P, Tsioulou P, Sfakianoudis K, Kontogeorgi A, Bakas P, Mastorakos G, Koutsilieris M, Simopoulou M. Investigating Stress Response during Vaginal Delivery and Elective Cesarean Section through Assessment of Levels of Cortisol, Interleukin 6 (IL-6), Growth Hormone (GH) and Insulin-Like Growth Factor 1 (IGF-1). J Clin Med. 2019 Jul 27;8(8):1112. doi: 10.3390/jcm8081112. PMID 31357604
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] Sultan P, Kamath N, Carvalho B, Bansal P, Elkhateb R, Dougan S, Whittington J, Guo N, El-Sayed Y, Mhyre J, Sharawi N. Evaluation of inpatient postpartum recovery using the Obstetric Quality of Recovery-10 patient-reported outcome measure: a single-center observational study. Am J Obstet Gynecol MFM. 2020 Nov;2(4):100202. doi: 10.1016/j.ajogmf.2020.100202. Epub 2020 Aug 17. PMID 33345919